CLINICAL TRIAL: NCT02779894
Title: Applicability, Efficacy and Cost Effectiveness of Sleep Apnoea Hypopnea Syndrome (SAHS) Management by an Information and Communication Based Technology (ICT)
Brief Title: Sleep Apnoea Management by a Communication Based Technology (ICT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Montserrat, Principal investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI14/00416
Record Dates: First submitted 2016-04-11; First posted 2016-05-23 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Obstructive Sleep Apnea; Telemedicine
Keywords: Sleep Apnea; Communication Based Technology; ICT
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hospital group (No Intervention): Patients referred to the sleep unit and randomized to Hospital group. Participants will be diagnosed in the hospital either by Polysomnography , Respiratory Polygraphy or one night Home Respiratory Polygraphy. In case of requiring CPAP treatment, the titration and adjustment of patient's will be accomplished at the hospital. This patient's will be monitored during 3 months of the study at the hospital.
- ICT group (Other): Patients referred to the sleep unit and randomized to intervention group. Participants will be diagnosed at home by 3 night Home Respiratory Polygraphy. In case of requiring CPAP treatment, the adjustment will be performed at the CPAP supplier center, titration will be performed at home and patient's compliance and treatment will be controlled via remote. During the 3 months of the study patient's will be controlled via phono/video conferences and with a platform designed for the study.
  Interventions: Other: Remote control of patients

INTERVENTIONS:
Other: Remote control of patients — Diagnosis outside the hospital (3 Home PR) CPAP (if needed) titration at home REmote control of patient's during 3 months by video or phonoconference
  Other Names: Communication based technology
  Arms: ICT group

SUMMARY:
This project develops a new form of management of subjects with suspected SAHS and different sleep disorders by applying Information and communications technologies (ICT).

DETAILED DESCRIPTION:
Sleep apnea hypopnea syndrome (SAHS) is a prevalent disease with significant morbidity resulting in long waiting lists and high health care costs. Therefore, alternative cost-effective approaches are urgently needed. A possible procedure is telemedicine based on ICT.

The design of the study is prospective, randomized, controlled, open and parallel.

A ICT-based out of hospital management of SAHS is implemented to be compared with the classical in-hospital management.

The main objectives were the evaluation of both groups and the analysis of efficacy and cost effectiveness of two SAHS management programs.

This is a 3 month randomized, with parallel groups study. Participants will be patients with suspicion of SAHS derived to the Investigators' Sleep Unit.

Patients are randomized in two groups; 1) classical in-hospital group: polysomnography or home respiratory polygraphy (HRP), CPAP titration and treatment and hospital follow-up; and 2) ICT group: 3 consecutive HRPs, automatic CPAP treatment and control by phone/video conferences and data transmission by using a custom designed platform.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of SAHS
* Use of Smartphone and internet

Exclusion Criteria:

* Severe hypersomnia
* Central apneas or other sleep disorder
* Previous CPAP treatment
* Unstable diseases
* Profession of risk
* Not able to complete questionnaires
* No written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the two SAHS management programs | 3 months
  Quebec sleep questionnaire
Evaluation of the two SAHS management programs | 3 months
  Compliance to CPAP treatment. (Number of hours that the patient uses CPAP)

SECONDARY OUTCOMES:
Cost-effectiveness of the two SAHS management programs | 3 months
  Costs of visits and transport of both groups (Bayesian analysis techniques)

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Montserrat, Study Director — Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes